CLINICAL TRIAL: NCT06797193
Title: Invoking Subharmonics and Subharmonic Aided Pressure Estimation (SHAPE) for Identifying Portal Hypertension
Brief Title: Ultrasound With Subharmonic Imaging and Subharmonic Aided Pressure Estimation (SHAPE) to Identify Portal Hypertension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Jaydev K. Dave, PhD, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-008738
Record Dates: First submitted 2025-01-22; First posted 2025-01-28 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Portal Hypertension
MeSH Terms: conditions — Hypertension, Portal | interventions — perflutren; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Diagnostic (Definity, SHAPE) (Experimental): Patients receive Definity IV once on study. Additionally, patients undergo ultrasound with and without SHAPE technique as well as standard of care liver biopsy on study.
  Interventions: Other: Electronic Health Record Review; Procedure: Liver Biopsy; Other: Medical Device Usage and Evaluation; Drug: Perflutren Lipid Microspheres; Procedure: Ultrasound Imaging

INTERVENTIONS:
Other: Electronic Health Record Review — Ancillary studies
Procedure: Liver Biopsy — Undergo liver biopsy
  Other Names: Biopsy of Liver
Other: Medical Device Usage and Evaluation — Undergo ultrasound with SHAPE technique
Drug: Perflutren Lipid Microspheres — Given IV
  Other Names: Definity
Procedure: Ultrasound Imaging — Undergo ultrasound
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasonography; Ultrasound; Ultrasound Test; Ultrasound, Medical; US

SUMMARY:
This clinical trial tests the how well an ultrasound with subharmonic imaging and the subharmonic aided pressure estimation (SHAPE) technique works in identifying portal hypertension (PH). An ultrasound takes pictures of the inside of the body by bouncing sound waves off organs. PH is high blood pressure in the vein that carries blood to the liver from the stomach, small and large intestines, spleen, pancreas, and gallbladder. The complications associated with PH are clear only after severe liver dysfunction or liver cirrhosis develops and are accompanied by relatively high mortality rates (20-70% mortality within 2 years). Thus, identifying PH earlier is beneficial. The hepatic venous pressure gradient (HVPG) obtained using an invasive catheterization procedure remains the standard for assessing PH. However, using this invasive procedure to assess PH prevents frequent pressure monitoring. Thus, a noninvasive technique to estimate PH is beneficial not only for diagnosis but also for monitoring treatment and disease progression. The SHAPE technique is a noninvasive ultrasound-based imaging technique that can estimate pressure with an ultrasound contrast agent. A noninvasive technique using an ultrasound with subharmonic imaging and the SHAPE technique may work in identifying PH.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate if SHAPE with perflutren lipid microspheres (Definity) microbubbles identifies patients with clinically significant PH.

II. To evaluate if addition of subharmonic imaging-based perfusion parameters derived from time intensity curves and shear wave elastography (SWE) measurements increase the diagnostic confidence of detecting PH.

OUTLINE:

Patients receive Definity intravenously (IV) once on study. Additionally, patients undergo ultrasound with and without SHAPE technique as well as standard of care liver biopsy on study.

After completion of study intervention, patients are followed up for 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated informed consent form
* Willing to comply with all study procedures
* Adult patients (age of 18 years or older)
* If a female of child-bearing potential, must have a negative pregnancy test
* Be scheduled for HVPG measurement

Exclusion Criteria:

* Patients who are unable to provide consent
* Females who are pregnant or nursing
* Patients with known or suspected hypersensitivity to perflutren lipid microsphere or its components, such as polyethylene glycol (PEG)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Clinically significant portal hypertension (PH) | Baseline (at time of ultrasound)
  Will evaluate if subharmonic aided pressure estimation with Definity microbubbles identifies patients with clinically significant PH.
Diagnostic confidence | Baseline (at time of ultrasound)
  Will evaluate if the addition of subharmonic imaging-based perfusion parameters increase the diagnostic confidence of detecting PH.

CONTACTS AND LOCATIONS:
Overall Officials: Jaydev K. Dave, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials